CLINICAL TRIAL: NCT05624359
Title: Flurbiprofen Axetil as an Adjuvant to Pre-emptive Scalp Infiltration for Post-craniotomy Pain
Brief Title: Flurbiprofen Axetil as an Adjuvant to Pre-emptive Scalp Infiltration
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: One case with postoperative subdural hematoma was reported to the Institutional Review Board and DMC. This study was suspended. The association with study interventions remained to be explored.
Sponsor: Beijing Tiantan Hospital (Other)
Responsible Party: Principal Investigator, Fang Luo, ProFessor, Beijing Tiantan Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2018-034-02-10
Record Dates: First submitted 2022-11-07; First posted 2022-11-22 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-09

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Ropivacaine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ropivacaine plus FA (Experimental): 5 mL FA (50 mg; by Beijing Taide Pharmaceutical Co., Ltd) and 15 mL of 1% ropivacaine (Nai Le Pin 10mg/mL; by AstraZeneca AB, Sweden) diluted to a total volume of 30 mL in normal saline
  Interventions: Drug: FA plus ropivacaine
- ropivacaine alone (Active Comparator): 15 mL of 1% ropivacaine diluted to a total volume of 30 mL in normal saline
  Interventions: Drug: ropivacaine alone

INTERVENTIONS:
Drug: FA plus ropivacaine — Th group will receive 0.17% FA and 0.5% ropivacaine for pre-emptive scalp infiltration at about 30 min before surgical incision. The assigned solution was injected along the planned surgical incision and pin fixation sites of the Mayfield head holder, using a 22-gauge needle introduced throughout the entire thickness of the scalp at a 45° angle.
  Arms: ropivacaine plus FA
Drug: ropivacaine alone — The ropivacaine alone group will receive 0.5% ropivacaine alone for pre-emptive scalp infiltration at about 30 min before surgical incision. The assigned solution was injected along the planned surgical incision and pin fixation sites of the Mayfield head holder, using a 22-gauge needle introduced throughout the entire thickness of the scalp at a 45° angle.
  Arms: ropivacaine alone

SUMMARY:
Post-craniotomy pain remains a major challenge in patient care following neurosurgery.Flurbiprofen axetil (FA), as an injectable nonselective cyclooxygenase inhibitor, is a widely prescribed NSAID for postoperative pain. As FA is highly lipophilic by merging into emulsified lipid microspheres, it has a high affinity to the surgical incision and inflammatory tissues to achieve targeted drug therapy and prolonged duration of action, thus providing a basis for its local use to achieve efficacy and safety comparable to or greater than systemic administration. In this study, we attempt to evaluate the clinical effects of FA as an adjunct to ropivacaine in pre-emptive scalp infiltration to prevent or reduce pain after craniotomy.

ELIGIBILITY:
Inclusion Criteria:

1. Age minimum 18 years;
2. ASA physical status of I - II;
3. Body mass index (BMI) of 15 - 30;
4. Scheduled for supratentorial craniotomy under general anesthesia;
5. Anticipated tracheal extubation, recovery of consciousness and orientation within 2 hours after craniotomy.

Exclusion Criteria:

1. Glasgow Coma Scale <15;
2. Unable to use the PCIA device or comprehend the pain NRS;
3. History of opioid dependence, chronic headache or intake of any drugs with known analgesic properties within the 24 hours before surgery;
4. History of craniotomy or scalp infection;
5. Any contraindication to flurbiprofen axetil, such as gastrointestinal ulcer, coagulation disorders, renal dysfunction, heart failure and ischemic heart disease;
6. History of allergy to any drug used in the study;
7. Pregnancy and breastfeeding.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 216 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Total consumption of sufentanil with PCIA device at 48 hours postoperatively. | at 48 hours postoperatively
  A postoperative Patient Controlled Intravenous Analgesia (PCIA) pump containing sufentanil 200μg in 100 mL saline will be administered from admission to the PACU until postoperative 48 hours.
  The PCIA pump will be set for 0.5 mL bolus doses with a lockout time of 15 min without initial dose or continuous infusion. The maximum dose will be limited to 2 mL (sufentanil 4 μg) per hour.

SECONDARY OUTCOMES:
Total consumption of sufentanil with PCIA pump at 24 hours after craniotomy | at 24 hours postoperatively
  A postoperative Patient Controlled Intravenous Analgesia (PCIA) pump containing sufentanil 200μg in 100 mL saline will be administered from admission to the PACU until postoperative 48 hours.
  The PCIA pump will be set for 0.5 mL bolus doses with a lockout time of 15 min without initial dose or continuous infusion. The maximum dose will be limited to 2 mL (sufentanil 4 μg) per hour.
Time to first PCIA button press after craniotomy | after craniotomy
  A postoperative Patient Controlled Intravenous Analgesia (PCIA) pump containing sufentanil 200μg in 100 mL saline will be administered from admission to the PACU until postoperative 48 hours.
  The PCIA pump will be set for 0.5 mL bolus doses with a lockout time of 15 min without initial dose or continuous infusion. The maximum dose will be limited to 2 mL (sufentanil 4 μg) per hour.
Pain NRS scores at 2 hours after craniotomy | at 2 hours after craniotomy
  0 indicates no pain and 10 indicates the worst pain imaginable
Pain NRS scores at 4 hours after craniotomy | at 4 hours after craniotomy
  0 indicates no pain and 10 indicates the worst pain imaginable
Pain NRS scores at 12 hours after craniotomy | at 12 hours after craniotomy
  0 indicates no pain and 10 indicates the worst pain imaginable
Pain NRS scores at 24 hours after craniotomy | at 24 hours after craniotomy
  0 indicates no pain and 10 indicates the worst pain imaginable
Pain NRS scores at 48 hours after craniotomy | at 48 hours after craniotomy
  0 indicates no pain and 10 indicates the worst pain imaginable
Pain NRS scores at 1 mon after craniotomy | at 1 mon after craniotomy
  0 indicates no pain and 10 indicates the worst pain imaginable
Pain NRS scores at 3 mons after craniotomy | at 3 mons after craniotomy
  0 indicates no pain and 10 indicates the worst pain imaginable
The time to first prescription of OC/APAP after craniotomy | up to 48 hours after craniotmy
  In the ward, if a patient scores > 4 in pain NRS after receiving a maximum dose of 2 mL per hour from PCIA device, an oral supplementary tablet of oxycodone (OC)/acetaminophen (APAP) (5/325 mg; by MallinckrodtInc, USA) will be prescribed as a rescue analgesic at an interval of at least 6 hours.
Hospital duration after craniotomy | From surgery day until the discharge date from hospital, assessed up to one week
  The duration from end of surgery to discharge from hospital
WHOQOL-BREF score | at 1month after craniotomy
  It is a questionnaire consisting of social relationships, physical health, psychological health, environment, overall QoL and general health. The mean score of each domain ranges between 4 and 20. A higher score indicates a better QoL
WHOQOL-BREF score | at 3 months after craniotomy
  It is a questionnaire consisting of social relationships, physical health, psychological health, environment, overall QoL and general health. The mean score of each domain ranges between 4 and 20. A higher score indicates a better QoL
PONV scores | at 24 hours after surgery
  It is rated as: 0, absent; 1, nausea not requiring treatment; 2, nausea requiring treatment; 3, vomiting
PONV scores | at 48 hours after surgery
  It is rated as: 0, absent; 1, nausea not requiring treatment; 2, nausea requiring treatment; 3, vomiting
Wound healing score | at 1 month after craniotomy
  It is rated as excellent, good and suboptimal
Wound healing score | at 3 months after craniotomy
  It is rated as excellent, good and suboptimal
Patient and Observer Scar Assessment Scale | at 1 month after craniotomy
  It consists of 2 numeric scales regarding the observer component (6 items) and the patient component (6 items). All included items are scored on the same 10-point scale. And a higher score represents a poorer scar quality.
Patient and Observer Scar Assessment Scale | at 3 months after craniotomy
  It consists of 2 numeric scales regarding the observer component (6 items) and the patient component (6 items). All included items are scored on the same 10-point scale. And a higher score represents a poorer scar quality.
The occurrence of other AEs | throughout both the treatment and follow-up periods (up to 3 months)
  Other AEs include cerebral hematoma, respiratory depression, gastrointestinal ulcerations and perforation, renal risks, coagulation dysfunction, allergic reaction and wound infection, oozing, hemorrhage, burning sensation and mild pruritus

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Tiantan Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No